CLINICAL TRIAL: NCT04357470
Title: Ulnar Styloid Fracture Accompanying Distal Radius Fracture Does Not Affect Functional Results, But What About Manual Dexterity?
Brief Title: Manual Dexterity in Ulnar Styloid Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, HANDE USTA, Principal Investigator, Research Assistant, Pamukkale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60116787020/62810
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Ulnar Styloid Fracture; Distal Radius Fracture
Keywords: DISTAL RADIUS FRACTURE; ULNAR STYLOID FRACTURE; MANUAL DEXTERITY
MeSH Terms: conditions — Wrist Fractures | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Patients who diagnosed diagnosed with isolated DRF or DRF accompanied with ulnar styloid fracture and applied to hand rehabilitation unit were included in the study. The patients were divided into two groups according to the ulnar styloid fracture presence. USF Group was DRF with ulnar styloid fracture; NON-USF Group was DRF without ulnar styloid fracture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- USF Group (Active Comparator): DRF with ulnar styloid fracture
  Interventions: Other: Hand Therapy
- NON-USF Group (Active Comparator): DRF without ulnar styloid fracture
  Interventions: Other: Hand Therapy

INTERVENTIONS:
Other: Hand Therapy — The patients were admitted to 12-weeks rehabilitation program and were called up once a week for follow-up appointments. Hand therapy continued as home program between 12th week and 6th month.
  Other Names: Rehabilitation

SUMMARY:
Fracture of the distal radius (DRF) is a common musculoskeletal system injury. Fracture of the ulnar styloid frequently accompanies fractures of the distal radius and is seen in 50-65% of these cases. The loss of dexterity is common in many musculoskeletal conditions.

The aim of this study was to investigate whether an associated ulnar styloid fracture following a distal radius fracture has any effect on manual dexterity.

Patients who diagnosed with isolated DRF or DRF accompanied with ulnar styloid fracture and applied to hand rehabilitation unit were included in the study. The patients were divided into two groups according to the ulnar styloid fracture presence. USF Group was DRF with ulnar styloid fracture; NON-USF Group was DRF without ulnar styloid fracture.

Pain, range of motion, Quick-DASH, hand grip and pinch strength, Purdue Pegboard Test, Jebsen Taylor Hand Function Test was measured at six month.

A total of 125 patients, 68 female (54,4%) and 57 male (45,6%) were included in the study. The mean age of the patients was 47,15±13,41 (18-65) years. 65 of the patients (52%) had isolated fracture of the distal radius fracture (NON-USF group) and 60 patients (48%) had a concurrent ulnar styloid fracture (USF group).

There was no significant difference in pain between the groups (p>0,05). Joints range of motion were higher in the NON-USF group than in the USF group. This difference was statistically significant only for flexion and extension (p<0,05). There was no statistically significant difference in Quick-DASH score between groups (p>0,05). The injured hand grip and pinch strength values in NON-USF group were greater than the USF group but the difference was not statistically significant (p>0,05). The manual dexterity and hand function tests showed that there was no statistically significant difference between the groups at six months (p>0,05).

There is a consensus that ulnar styloid fracture has no effect on overall hand function. But, there is no study dwelled on the manual dexterity. In this study, the effect of ulnar styloid fracture on hand function is more clearly emphasized. In conclusion, concomitant USF does not lead poorer manual dexterity.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for inclusion in this prospective cohort study were; 1) Aged between 18 and 60 years, 2) Diagnosed with isolated DRF or DRF accompanied with ulnar styloid fracture, 3) Primarily fixation after injury

Exclusion Criteria:

* Exclusion criteria were; 1)Radius shaft, ulnar head or ulnar shaft fractures, 2) Pre-existing rheumatological diseases associated with ipsilateral extremity, 3) Comorbid injuries such as tendon or nerve injuries, 4) Coexisting distal radioulnar, radiocarpal or ulnocarpal joint instability problems, 5) Secondarily repair.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2019-09-14 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Pain | six month
  The severity of pain was assessed with a visual analogue scale (VAS) in sleep, rest, and activity
Range of motion | six month
  Patients' forearm and wrist joints ROM (pronation, supination, flexion, extension, radial and ulnar deviation) were measured with an universal goniometer
Grip and Pinch Strength | six month
  The handgrip and pinch strengths were measured according to standard strength measurement method suggested by American Society of Hand Therapists respectively using a hand dynamometer and a pinch meter
Quick-The Disabilities of the Arm, Shoulder and Hand (Q-DASH) | six month
  It was used to a shortened version of the DASH Outcome Measure. Instead of 30 items, the Quick-DASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb
Purdue Pegboard Test | six month
  Four subtests of the Purdue Pegboard Test (1-800-428-7545, Model 32020, Lafayette Instrument Co., IL, USA) (right hand, left hand, both hands and assembly) were performed to measure fine manual dexterity of the hands after DRF
Jebsen Taylor Hand Function Test | six month
  The seven individual subtests of JTHFT (Sammons Preston Ability One, #8063) including writing, card turning, picking up small common objects, stacking checkers, stimulated feeding, moving light objects and moving heavy objects were performed in a standardized procedure

CONTACTS AND LOCATIONS:
Overall Officials: HANDE USTA, MSC, Principal Investigator — Research Assistant

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almedghio S, Arshad MS, Almari F, Chakrabarti I. Effects of Ulnar Styloid Fractures on Unstable Distal Radius Fracture Outcomes: A Systematic Review of Comparative Studies. J Wrist Surg. 2018 Apr;7(2):172-181. doi: 10.1055/s-0037-1607214. Epub 2017 Oct 11. PMID 29576925
- [Background] Yuan C, Zhang H, Liu H, Gu J. Does concomitant ulnar styloid fracture and distal radius fracture portend poorer outcomes? A meta-analysis of comparative studies. Injury. 2017 Nov;48(11):2575-2581. doi: 10.1016/j.injury.2017.08.061. Epub 2017 Aug 31. PMID 28882374
- [Background] Yong J, MacDermid JC, Packham T. Defining dexterity-Untangling the discourse in clinical practice. J Hand Ther. 2020 Oct-Dec;33(4):517-519. doi: 10.1016/j.jht.2019.11.001. Epub 2020 Jan 16. No abstract available. PMID 31956020